CLINICAL TRIAL: NCT02193763
Title: Bedside Ultrasound Assisted Pediatric Lumbar Puncture--A Randomized Controlled Trial
Brief Title: Bedside Ultrasound Assisted Pediatric Lumbar Puncture
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has relocated to another institution, no other site PI to take over
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AHC 4746
Record Dates: First submitted 2014-07-13; First posted 2014-07-18 (Estimated); Last update posted 2024-10-04 (Actual); Status verified 2024-06

CONDITIONS: Infant/ Neonate Lumbar Puncture
Keywords: pediatric; lumbar puncture; ultrasonography; efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 90 days and under--Interventional (Experimental): Neonates aged 90 days and under randomized to ultrasound assisted lumbar puncture
  Interventions: Procedure: Ultrasound assisted lumbar puncture
- 90 days and under--control (No Intervention): Neonates aged 90 days and under randomized to lumbar puncture using the anatomical landmark approach
- Over 90 days--Interventional (Experimental): Neonates aged over 90 days randomized to ultrasound assisted lumbar puncture
  Interventions: Procedure: Ultrasound assisted lumbar puncture
- Over 90 days--Control (No Intervention): Neonates aged over 90 days randomized to lumbar puncture using the anatomical landmark approach

INTERVENTIONS:
Procedure: Ultrasound assisted lumbar puncture — An investigator will perform beside ultrasound on the spinal area using a bedside ultrasound device. Attempts will be made to visualize the spinous processes and vertebral bodies in the general lumbarsacral area, as well as the presence of CSF in the thecal space below the conus medullaris, and identify the optimal location to perform the LP. This will be marked with a skin marker (If no CSF or abnormal anatomy is visualized, the LP will be advised to be postponed or cancelled). The treating physician will then proceed with the LP guided by the skin markings.
  Other Names: Sonosite M-Turbo ultrasound device (Bothell, WA) with a L25 linear transducer; or; Zonare Z.One device(Mountain View, CA) with a L10-5 linear array transducer,
  Arms: 90 days and under--Interventional; Over 90 days--Interventional

SUMMARY:
This is a prospective, randomized study evaluating the efficacy of bedside ultrasound assisted lumbar puncture in pediatric patients

DETAILED DESCRIPTION:
Comparison of bedside ultrasound assisted lumbar puncture to traditional anatomical landmark approach in neonates and young infants requiring lumbar puncture

ELIGIBILITY:
Inclusion Criteria:

* Any patient 0-12 months old requiring a lumbar puncture in the pediatric emergency department or inpatient pediatric floor is eligible to participate in the study

Exclusion Criteria:

* previous back surgeries
* parent/ guardian inability to understand informed consent
* parent/guardian refusal of informed consent.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2024-06 (Actual); Study Completion 2024-06 (Actual)

PRIMARY OUTCOMES:
Traumatic lumbar puncture | up to 24 hours
  RBC>10,000/ mm3 on spinal fluid analysis
Unsuccessful lumbar puncture | average of <1hour
  failure to yield enough fluid for cerebrospinal fluid cell count as indicated by operator report on data collection sheet

SECONDARY OUTCOMES:
Hospital length of stay | average of <7days
  as reported in the subjects' medical record

OTHER OUTCOMES:
clinical outcome/ hospital course of the patient | 30days
  whether there was any adverse effect/ complication due to lumbar puncture based on review of medical record
number of lumbar puncture attempts | average of <1hour
  as recorded on the data collection form
time to completion of lumbar puncture | average of <1hour
  as reported in the data collection form (measured in seconds)
perception of the clinician on the usefulness of bedside ultrasound if used | up to 24 hours
  as rated on a 1-5 Likert scale by the operator on the data collection form

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Lam, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Advocate Christ Medical Center, Oak Lawn, Illinois, United States